CLINICAL TRIAL: NCT02682173
Title: MRI Fat Quantification of the Liver, Subcutaneous and Visceral Fatty Tissue in Patients Before and After Bariatric Surgery
Brief Title: Magnetic Resonance Imaging (MRI) Fat Quantification of the Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MRI Fat quantification
Record Dates: First submitted 2016-02-01; First posted 2016-02-15 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Non-alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic gastric bypass (Active Comparator): MR Abdomen in morbidly obese patients receiving gastric bypass
  Interventions: Other: MR Abdomen
- Laparoscopic sleeve gastrectomy (Active Comparator): MR Abdomen morbidly obese patients receiving sleeve gastrectomy
  Interventions: Other: MR Abdomen

INTERVENTIONS:
Other: MR Abdomen

SUMMARY:
Fatty liver in the obese is a common finding; some cases develop steato-hepatosis which in the long-term can lead to liver cirrhosis. The effect of bariatric surgery on fat distribution in the liver has so far been studied with liver biopsies and single voxel MR techniques. With this trial investigators present a new, whole organ MR-quantification of liver fat and describe changes after bariatric surgery in visceral and subcutaneous fat.

DETAILED DESCRIPTION:
Currently, liver biopsy is still regarded as the gold-standard in the diagnosis of non-alcoholic fatty liver disease and monitoring of progression. However, accuracy of diagnosis is not perfect with a certain risk of sampling error depending on biopsy quality and a more or less homogeneous distribution of liver tissue alterations. Complications are rare; however, the method is invasive and carries the risk of bleeding. Therefore, non-invasive methods (such as serum biomarkers or imaging techniques) are sought for accurate diagnosis and safe monitoring of disease progression. Unidimensional transient elastography (TE; FibroScan®) is a non-invasive technique, which can be a helpful tool here: however, accuracy of diagnosis is depending on the stage of fibrosis and lower grades of fibrosis (stage 1 and 2) are difficult to assess. Moreover, in obese patients this method cannot be applied.

In recent years, the development of fat-water magnetic resonance imaging has enabled non-invasive assessment of fat and water content in tissues. In addition, modern MRI devices allow brief breath holding, which reduces motion artifacts and provides us with excellent data and therefore MRI has become an important tool for fat quantification.

Up to date only a few studies have focused on fat quantification before and after bariatric surgery: patients treated with laparoscopic gastric banding (a purely restrictive procedure) and patients undergoing metabolic surgery such as sleeve gastrectomy and gastric bypass have been examined pre- and postoperatively by means of MRI fat quantification. However, in these studies single voxel spectroscopy was used. In contrast, in this current trial investigators aim to assess full organ volume, which hopefully will provide more accurate data.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients with BMI over 35, scheduled for bariatric surgery (either sleeve gastrectomy or gastric bypass)

Exclusion Criteria:

* Smoking
* substance abuse
* Diabetes
* history of gastrointestinal disorders
* pace-maker
* claustrophobia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Liver fat quantification | within 3, 6 and 12 months of surgery
  change in fat quantification; measurement of fat rate in the organ

SECONDARY OUTCOMES:
Visceral fat quantification | within 3, 6 and 12 months of surgery
  change in fat quantification visceral; 2-point Dixon technique for volumetric fat imaging
Subcutaneous fat quantification | within 3, 6 and 12 months of surgery
  change in fat quantification subcutaneous; 2-point Dixon technique for volumetric fat imaging

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer-Gerspach AC, Peterli R, Moor M, Madorin P, Schotzau A, Nabers D, Borgwardt S, Beglinger C, Bieri O, Wolnerhanssen BK. Quantification of Liver, Subcutaneous, and Visceral Adipose Tissues by MRI Before and After Bariatric Surgery. Obes Surg. 2019 Sep;29(9):2795-2805. doi: 10.1007/s11695-019-03897-2. PMID 31089967